CLINICAL TRIAL: NCT06013592
Title: Gut Hormone LEAP2 in Metabolism and Eating Behaviour: Fixed Meal Testing
Acronym: LEAP2-meal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 23HH8298
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Eating Behavior; Obesity; Appetitive Behavior
Keywords: LEAP2; ghrelin; appetite; food intake; eating behaviour
MeSH Terms: conditions — Feeding Behavior; Obesity; Appetitive Behavior | interventions — Single Person; Population Groups; Adiposity

STUDY DESIGN:
Intervention Model Description: within participant
Who Masked: Participant
Masking Description: single-blinded, randomized order
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy adults without obesity (Experimental): Liquid meals with different caloric sizes (0, 600, 900, 1200 kcal) in within-participant cross-over design
  Interventions: Dietary Supplement: 0 kcal liquid meal; Dietary Supplement: 600 kcal liquid meal; Dietary Supplement: 900 kcal liquid meal (only for group without obesity); Dietary Supplement: 1200 kcal liquid meal
- Healthy adults with obesity (Experimental): Liquid meals with different caloric sizes (0, 600, 1200, 1800 kcal) in within-participant cross-over design
  Interventions: Dietary Supplement: 0 kcal liquid meal; Dietary Supplement: 600 kcal liquid meal; Dietary Supplement: 1200 kcal liquid meal; Dietary Supplement: 1800 kcal liquid meal (only for group with obesity)

INTERVENTIONS:
Dietary Supplement: 0 kcal liquid meal — Flavoured water, given as one meal at one study visit only
Dietary Supplement: 600 kcal liquid meal — Fortisip Compact Vanilla, given as one meal at one study visit only
Dietary Supplement: 900 kcal liquid meal (only for group without obesity) — Fortisip Compact Vanilla, given as one meal at one study visit only
  Arms: Healthy adults without obesity
Dietary Supplement: 1200 kcal liquid meal — Fortisip Compact Vanilla, given as one meal at one study visit only
Dietary Supplement: 1800 kcal liquid meal (only for group with obesity) — Fortisip Compact Vanilla, given as one meal at one study visit only
  Arms: Healthy adults with obesity

SUMMARY:
The goal of this interventional study is to measure the blood levels of the gut hormones LEAP2 and acyl ghrelin (AG), appetite and food intake after consuming liquid meals of different caloric sizes, in healthy adults with and without obesity.

AG is a stomach-derived homone that increases appetite, and LEAP2 a liver-gut derived hormone that decreases appetite, which interferes the action of AG ant its receptor in the brain called the growth hormone secretagogue receptor (GHSR). Blood levels of AG and LEAP2 change in opposite directions after food intake (AG decreasing, LEAP2 increasing). AG is formed from an inactive version of hormone called desacyl ghrelin (DAG). Previous studies have shown that greater food intake leads to a greater decrease in blood levels of total ghrelin (AG + DAG), but this has not been studied for changes in blood AG or LEAP2 after eating. Blood levels of AG and total ghrelin when fasted and after food intake are lower, while blood levels of LEAP2 are higher, in adults with than those without obesity.

The main study questions are:

1. Are there greater increases in blood levels of LEAP2 and greater decreases in blood levels of AG after consuming larger meals (by amount of calories they contain)?
2. Are greater decreases in appetite after connsuming larger meals related to greater increases in blood levels of LEAP2 and greater decreases in blood levels of AG?
3. Are greater decreases in food intake at a buffet lunch after consuming larger meals eaten a few hours previously related to greater increases in blood levels of LEAP2 and greater decreases in blood levels of AG?
4. Do the above findings differ between adults without obesity and with obesity?

At each of 4 study days, healthy adults (without and with obesity) will consume one size of a single liquid meal containing different amounts of calories (0, 600, 900 (group without obesity only), 1200, 1800 (group with obesity only) kilocalories, of identical total volume) after an overnight fast and have measurements of blood LEAP2 and AG and appetite ratings from 0 to 180 min, and have food intake at an ad libitum lunch measured at 180 mins. Food will be weighed and converted into kilocalories.

All participants will attend for all 4 study visits in a randomised order to receive one of the meal sizes at each visit, so that all 4 meal zizes are consumed over all 4 study visits: 0, 600, 900 (group without obesity), 1200, 1800 (group with obesity) kcal.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 60 years;
* Without obesity with body mass index (BMI) 18.0-29.9 kg/m2 or with obesity with BMI 30.0-50.0 kg/m2;
* Healthy as determined by medical history and vital signs;
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form;
* Participant is able to read, comprehend and record information written in English.

Exclusion Criteria:

* History of, or current abuse or dependence on alcohol or drugs;
* Current smoker or less than 2 years since quitting (cigarette, cigars, e-cigarettes) or use of nicotine replacement therapy;
* Significant current or past medical or psychiatric history that, in the opinion of the investigators, contraindicates their participation;
* History of type 1 or type 2 diabetes mellitus;
* History of ischaemic heart disease, heart failure, cardiac arrhythmia, peripheral vascular, cerebrovascular disease or uncontrolled hypertension;
* Current diagnosis of anaemia or iron deficiency;
* Body weight instability (change in body weight of more than 5% over the preceding 3 months);
* Use of current regular prescription or over-the-counter medications that in the opinion of the Investigators may affect participant safety or outcome measures;
* Clinically significant abnormalities in screening blood tests abnormalities which in the opinion of the study physician, is clinically significant e.g. diabetes mellitus, hypothyroidism, renal impairment, abnormal liver function tests [bilirubin, alanine transaminase (ALT), aspartate transaminase (AST), gamma-glutamyl transferase (GGT)] >3x upper limit of normal, other than due to fatty liver disease; Current pregnancy or breast-feeding in female volunteers (the Investigators will recommend using contraception for the duration of the visits to avoid participant drop-out);
* Pulse rate <40 or >100 beats per minute OR systolic blood pressure >160 and <100 OR diastolic blood pressure >95 and <50 in the semi-supine position;
* Volunteer has participated in a clinical trial and has received an investigational product within the following time period prior to the first experimental visit in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer);
* Exposure to more than 3 new investigational medicinal products within 12 months prior to the scan;
* Vegan, gluten or lactose-intolerant (as test meals in the paradigms may include animal products, dairy and wheat products);
* Volunteers who have donated, or intend to donate, blood within three months before the screening visit or following study visit completion;
* Known history of SARS-CoV-2 infection (Covid-19) in the last 4 weeks;
* Ongoing symptoms suggestive of complications from previous SARS-CoV-2 infection ('long Covid-19') such as loss or change in sense of smell or taste, shortness of breath, palpitations, lethargy;
* SCOFF questionnaire score >1/5 indicating eating disorders (Luck et al. 2002);
* DSM-V criteria for alcohol use disorder (AUD) >2/11 indicating mild AUD (American-Psychiatric-Association 2013);
* Participants who have had previous obesity surgery or are on medications for obesity;
* Dutch Eating Behaviour Questionnaire (DEBQ) restraint score >3/5 indicating highly restrained eating behaviour.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Post-prandial plasma concentration acyl ghrelin | 0, 30, 60, 120, 180 minutes
  Incremental area under curve (iAUC) 0-180 minutes, units: pg/mL.hr
Post-prandial plasma concentration LEAP2 | 0, 30, 60, 120, 180 minutes
  Incremental area under curve (iAUC) 0-180 minutes, units: ng/mL.hr

SECONDARY OUTCOMES:
Visual analogue scale ratings of appetite | 0, 30, 60, 120, 180 minutes
  Incremental area under curve (iAUC) 0-180 minutes - units: mm.hr
Ad libitum food intake | at 180 minutes
  Total kilocalories eaten as % estimated resting energy expenditure (calculated from bio-impedance analysis determined fat free mass using Cunningham equation equating with lean body mass)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Goldstone, MRCP PhD, Principal Investigator — Imperial College London
Locations (1):
- PsychoNeuroEndocrinology Research Group, Division of Psychiatry, Dept. of Brain Sciences, Imperial College London, London, United Kingdom